CLINICAL TRIAL: NCT02640547
Title: Real World Evidence (RWE) of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Poland (HCV RWE PMOS)
Brief Title: Real World Evidence of the Effectiveness of Paritaprevir/Ritonavir, Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: IST GmbH, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-767; PLHCVRWE01 (Other Grant/Funding Number: Affiliate Study Tracking Number)
Record Dates: First submitted 2015-12-21; First posted 2015-12-29 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Dasabuvir; Paritaprevir/r/Ombitasvir; Observational Study; Quality of Life; Fibrosis; Cirrhosis; Work Ability
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin: Participants in this observational study received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
  The prescription of treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
This study seeks to provide evidence of the effectiveness and obtain patient reported outcomes (PRO) and work productivity data of the interferon-free regimen of paritaprevir (PTV)/ritonavir (r) + ombitasvir (OBV), +/- dasabuvir (DSV), +/- ribavirin (RBV) in chronic hepatitis C virus infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female patients with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with the current local label.
* If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy).
* Patients must voluntarily sign and date a patient authorization to use and/or disclose his/her anonymized health data prior to inclusion into the study.
* Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

-None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis C (CHC)
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this prospective, multi-center observational study a total of 394 adult patients chronically infected with hepatitis C virus (HCV) were enrolled at 17 centers in Poland.
Pre-assignment Details: Effectiveness analyses of clinical outcomes are reported by HCV genotype. Safety variables were analyzed by treatment regimen.
Period: Overall Study
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Started | 394
Completed (HCV ribonucleic acid (RNA) treatment assessment performed at least 10 weeks post-treatment) | 383
Not Completed | 11
Not completed — Failure to Return | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 6
Not completed — Miscellaneous | 3

BASELINE CHARACTERISTICS:
Arm/Group | Paritaprevir/Ritonavir + Ombitasvir ± Dasabuvir ± Ribavirin
Number analyzed (Participants) | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 316
  66 to 84 years | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 394
Years Since Diagnosis of HCV Infection [Mean (Standard Deviation); unit: years] | 6.6 (5.94)
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1a | 24
  Genotype 1a/1b | 1
  Genotype 1b | 349
  Genotype 4 | 20
Cirrhosis Status [Count of Participants; unit: Participants]
  No cirrhosis | 211
  Transition to cirrhosis | 58
  Cirrhosis | 125

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: Enrolled participants who received adequate treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) according to standard of care and within local label recommendations for their specific disease characteristics.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Genotype 1 (Total): Participants with genotype 1 HCV received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
- Genotype 1a: Participants with genotype 1a HCV received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
- Genotype 1b: Participants with genotype 1b HCV received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
- Genotype 4: Participants with genotype 4 HCV received treatment with paritaprevir/ritonavir (r) and ombitasvir with or without dasabuvir ± ribavirin (RBV) for 12 or 24 weeks for the treatment of chronic hepatitis C (CHC), according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease.
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
percentage of participants | 96.8 [94.5 to 98.2] | 100.0 [86.7 to 100.0] | 96.6 [94.1 to 98.0] | 95.0 [76.4 to 99.1]

2. Secondary Outcome: Percentage of Participants Achieving Virological Response at End of Treatment
Description: Virologic response is defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen)
Population: Enrolled participants who received adequate treatment with paritaprevir/r and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin according to standard of care and within local label recommendations for their specific disease characteristics.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
percentage of participants | 95.5 [92.8 to 97.1] | 100.0 [86.7 to 100.0] | 95.1 [92.3 to 96.9] | 100.0 [83.9 to 100.0]

3. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as participants with a virologic response (VR; HCV RNA < 50 IU/mL) at end of treatment (EOT) followed by HCV RNA ≥ 50 IU/mL at any time after the end of treatment.
Time Frame: End of treatment (week 12 or 24 depending on the treatment regimen) and up to 24 weeks after the end of treatment.
Population: Participants who received adequate treatment with the ABBVIE REGIMEN ± RBV according to standard of care and within local label recommendations for their specific disease characteristics, and with VR at actual EOT and who completed treatment, and had ≥ 1 HCV RNA measurement ≥ 70 days post-treatment or were a treatment failure between EOT and day 70
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 349 | 25 | 324 | 19
percentage of participants | 0.6 [0.2 to 2.1] | 0.0 [0.0 to 13.3] | 0.6 [0.2 to 2.2] | 0.0 [0.0 to 16.8]

4. Secondary Outcome: Percentage of Participants With Breakthrough
Description: Breakthrough was defined as at least one documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: 12 or 24 weeks (depending on the treatment regimen)
Population: Participants who received adequate treatment with the ABBVIE REGIMEN ± RBV according to standard of care and within local label recommendations for their specific disease characteristics, who had at least one undetectable HCV RNA measurement on-treatment and at least one measurement on-treatment thereafter
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 17 | 1 | 16 | 5
percentage of participants | 0.0 [0.0 to 18.4] | 0.0 [0.0 to 79.3] | 0.0 [0.0 to 19.4] | 0.0 [0.0 to 43.4]

5. Secondary Outcome: Percentage of Participants With a Rapid Virological Response at Week 4
Description: Rapid virological response at week 4 (RVR4) was defined as participants with HCV RNA < 50 IU/mL at week 4.
  Due to the non-interventional character of the study, many participants did not have an HCV RNA assessed at treatment week 4 since this is not generally recommended in the label. Participants with missing data at the RVR4 time point were considered as virological failures.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
percentage of participants | 3.7 [2.2 to 6.2] | 0.0 [0.0 to 13.3] | 4.0 [2.4 to 6.6] | 5.0 [0.9 to 23.6]

6. Secondary Outcome: Percentage of Participants Achieving Sustained Virological Response 24 Weeks Post-treatment (SVR24)
Description: Sustained virologic response is defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 24 weeks after the last dose of study drug.
Time Frame: 24 weeks after the last dose of study drug (week 36 or 48 depending on the treatment regimen)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
percentage of participants | 96.3 [93.8 to 97.8] | 100.0 [86.7 to 100.0] | 96.0 [93.4 to 97.6] | 95.0 [76.4 to 99.1]

7. Secondary Outcome: Percentage of Participants in the Core Population With Sufficient Follow-up Data for SVR12 Who Achieved Sustained Virological Response 12 Weeks Post-treatment (SVR12)
Description: Sustained virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) levels less than 50 IU/mL 12 weeks after the last dose of study drug.
  The core population with sufficient follow-up data regarding SVR12 included all core population participants who
  * had evaluable HCV RNA data ≥ 70 days after the last actual dose of the ABBVIE regimen,
  * or a HCV RNA value ≥ 50 IU/mL at the last measurement post-baseline
  * or had HCV RNA < 50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥ 70 days after the last actual dose of the ABBVIE regimen due to reasons related to safety (e.g. dropped out due to adverse event) or virologic failure.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: The core population with sufficient follow-up data regarding SVR12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 371 | 25 | 346 | 20
percentage of participants | 97.6 [95.5 to 98.7] | 100.0 [86.7 to 100.0] | 97.4 [95.1 to 98.6] | 95.0 [76.4 to 99.1]

8. Secondary Outcome: Percentage of Participants in Each Non-response Category 12 Weeks Post-treatment
Description: SVR12 non-response was categorized according to the following:
  * Relapse, defined as HCV RNA < 50 IU/mL at EOT followed by HCV RNA ≥ 50 IU/mL post-treatment in patients who completed treatment (not more than 7 days shortened);
  * Death;
  * Premature treatment discontinuation with no on-treatment virological failure;
  * Missing SVR12 data and/or none of the above criteria.
Time Frame: 12 weeks after the last dose of study drug (week 24 or 36 depending on the treatment regimen)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
percentage of participants
  Relapse | 0.5 | 0.0 | 0.6 | 0.0
  Death | 1.6 | 0.0 | 1.7 | 0.0
  Premature treatment discontinuation | 0.3 | 0.0 | 0.3 | 5.0
  Missing SVR12 data/None of the above | 0.8 | 0.0 | 0.9 | 0.0

9. Secondary Outcome: Assigned Treatment Regimen
Description: Treatment regimen was assigned by the physician according to local practice and label. Participants could receive two direct-acting antiviral (DAA) drugs (paritaprevir/ritonavir and ombitasvir) plus ribavirin (RBV) for either 12 or 24 weeks, or three DAAs (paritaprevir/ritonavir, ombitasvir, and dasabuvir) with or without RBV for 12 or 24 weeks.
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
Participants
  2 DAA + RBV (12 weeks) | 0 | 0 | 0 | 8
  2 DAA + RBV (24 weeks) | 0 | 0 | 0 | 11
  3 DAA without RBV (12 weeks) | 229 | 0 | 229 | 0
  3 DAA + RBV (12 weeks) | 141 | 22 | 119 | 1
  3 DAA + RBV (24 weeks) | 4 | 3 | 1 | 0

10. Secondary Outcome: Percentage of the Direct Acting Antiviral (DAA) Dose Taken in Relation to the Target Dose of DAA
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: All enrolled participants who received at least one dose of the ABBVIE REGIMEN.
Measure: Count of Participants; unit: Participants
Groups:
- 2 DAA + RBV: Participants received paritaprevir/ritonavir and ombitasvir plus ribavirin for either 12 or 24 weeks.
- 3 DAA Without RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir without RBV for 12 weeks.
- 3 DAA + RBV: Participants received paritaprevir/ritonavir, ombitasvir, and dasabuvir with ribavirin for 12 or 24 weeks.
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 229 | 146
Participants
  > 95% | 18 | 227 | 141
  > 80 % to ≤ 95% | 0 | 0 | 1
  > 50% to ≤ 80% | 0 | 1 | 2
  ≤ 50% | 1 | 1 | 2

11. Secondary Outcome: Percentage of the Ribavirin (RBV) Dose Taken in Relation to the Target Dose of RBV
Description: Adherence to study treatment was calculated as:
  Cumulative dose taken / (initial prescribed dose * planned duration)
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: All enrolled participants who received at least one dose of the ABBVIE REGIMEN that included ribavirin
Measure: Count of Participants; unit: Participants
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 0 | 146
Participants
  > 95% | 14 |  | 105
  > 80% to ≤ 95% | 1 |  | 8
  > 50% to ≤ 80% | 0 |  | 19
  ≤ 50% | 4 |  | 14

12. Secondary Outcome: Number of Participants With Comorbidities
Time Frame: Baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype 1 (Total) | Genotype 1a | Genotype 1b | Genotype 4
Number analyzed (Participants) | 374 | 25 | 349 | 20
Participants
  Any comorbidity or coinfection | 224 | 10 | 214 | 16
  Any coinfection | 15 | 2 | 13 | 4
  Coinfection with human immunodeficiency virus (HIV | 8 | 2 | 6 | 4
  Coinfection with hepatitis B virus | 8 | 0 | 8 | 0

13. Secondary Outcome: Number of Participants Who Received Concomitant Medications
Description: Concomitant medication other than for chromic hepatitis C used from the time when the decision was made to initiate treatment with the ABBVIE REGIMEN until after the last dose.
Time Frame: From first dose of study drug to end of treatment, 12 to 24 weeks depending on the treatment regimen
Population: All enrolled participants who received at least one dose of the ABBVIE REGIMEN.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 229 | 146
Participants | 10 | 103 | 64

14. Secondary Outcome: Number of Participants With Adverse Events, Serious Adverse Events, or Pregnancies
Time Frame: From first dose of study drug through 30 days after last dose. The median duration of treatment was 84 days.
Population: All enrolled participants who received at least one dose of the ABBVIE REGIMEN.
Measure: Count of Participants; unit: Participants
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 229 | 146
Participants
  Any adverse event | 8 | 19 | 42
  Serious adverse events | 3 | 3 | 8
  Pregnancies | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. The 5 items in the EQ-5D-5L comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate visual analog scale (VAS).
  Responses to the 5 dimension scores were combined and converted into a single preference-weighted health utility index score by applying country-specific weights.The range for EQ-5D-5L index score is 0 to 1 where '0' is defined as a health state equivalent to being dead and '1' is full health.The higher the score the better the health status.
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks after end of treatment
Population: Enrolled participants who received adequate treatment with paritaprevir/r and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) according to standard of care and within local label recommendations for their specific disease characteristics. Participants with available data at baseline and each time point are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 221 | 139
units on a scale
  End of treatment: number analyzed (Participants) | 19 | 218 | 135
  End of treatment | 0.06 [0.01 to 0.10] | 0.04 [0.03 to 0.06] | 0.04 [0.02 to 0.06]
  12 weeks post treatment: number analyzed (Participants) | 18 | 217 | 134
  12 weeks post treatment | 0.07 [0.02 to 0.11] | 0.05 [0.04 to 0.07] | 0.04 [0.02 to 0.06]
  24 weeks post treatment: number analyzed (Participants) | 18 | 218 | 132
  24 weeks post treatment | 0.05 [-0.00 to 0.11] | 0.07 [0.05 to 0.08] | 0.04 [0.02 to 0.06]

16. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension 5 Level (EQ-5D-5L) VAS Score
Description: The EQ-5D-5L is a health state utility instrument that evaluates preference for health status. with a separate visual analog scale (VAS).
  The VAS assesses overall health on a scale from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks after end of treatment
Population: Enrolled participants who received adequate treatment with paritaprevir/r and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± RBV according to standard of care and within local label recommendations for their specific disease characteristics. Participants with available data at baseline and each time point are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 229 | 146
units on a scale
  End of treatment: number analyzed (Participants) | 19 | 227 | 143
  End of treatment | 4.10 [-1.52 to 9.73] | 7.41 [5.79 to 9.04] | 5.13 [3.08 to 7.17]
  12 weeks post treatment: number analyzed (Participants) | 18 | 227 | 142
  12 weeks post treatment | 7.93 [1.90 to 14.0] | 9.11 [7.41 to 10.8] | 7.01 [4.86 to 9.15]
  24 weeks post treatment: number analyzed (Participants) | 18 | 225 | 139
  24 weeks post treatment | 6.54 [0.74 to 12.3] | 11.8 [10.2 to 13.4] | 9.20 [7.11 to 11.3]

17. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Absenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Absenteeism indicates the percentage of work time missed due to health problems.
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks post treatment
Population: Enrolled participants who received adequate treatment with paritaprevir/r and ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± RBV according to standard of care and within local label recommendations for their specific disease characteristics. Participants who were employed with available data at baseline and each time point are included.
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 9 | 87 | 43
percent impairment
  End of treatment: number analyzed (Participants) | 6 | 80 | 35
  End of treatment | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  12 weeks post treatment: number analyzed (Participants) | 4 | 81 | 38
  12 weeks post treatment | 0.0 [-11.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.]
  24 weeks post treatment: number analyzed (Participants) | 5 | 77 | 36
  24 weeks post treatment | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

18. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Presenteeism
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Presenteeism indicates the percentage of impairment while working due to health problems.
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks after end of treatment
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 9 | 88 | 44
percent impairment
  End of treatment: number analyzed (Participants) | 6 | 79 | 34
  End of treatment | -5.0 [-10.0 to 10.0] | 0.0 [-20.0 to 0.0] | 0.0 [-10.0 to 0.0]
  12 weeks post treatment: number analyzed (Participants) | 4 | 79 | 39
  12 weeks post treatment | -5.0 [-20.0 to 0.0] | 0.0 [-20.0 to 0.0] | 0.0 [-10.0 to 0.0]
  24 weeks post treatment: number analyzed (Participants) | 5 | 76 | 37
  24 weeks post treatment | -10.0 [-20.0 to 0.0] | -10.0 [-20.0 to 0.0] | 0.0 [-20.0 to 0.0]

19. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Work Productivity Impairment (TWP)
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment (TWP) indicates the percentage of overall work impairment due to health problems.
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks after end of treatment
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 9 | 87 | 43
percent impairment
  End of treatment: number analyzed (Participants) | 6 | 80 | 35
  End of treatment | -5.0 [-10.0 to 10.0] | 0.0 [-20.0 to 0.0] | 0.0 [-10.0 to 0.0]
  12 weeks post treatment: number analyzed (Participants) | 4 | 79 | 38
  12 weeks post treatment | -5.0 [-27.7 to 0.0] | 0.0 [-20.0 to 0.0] | 0.0 [-10.0 to 0.0]
  24 weeks post treatment: number analyzed (Participants) | 5 | 77 | 36
  24 weeks post treatment | -10.0 [-20.0 to 0.0] | -10.0 [-20.0 to 0.0] | 0.0 [-20.0 to 0.0]

20. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI): Total Activity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment (TAI) indicates the percentage of general (non-work) activity impairment due to health problems.
Time Frame: Baseline, end of treatment, and at 12 and 24 weeks after end of treatment
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: percent impairment
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
Number analyzed (Participants) | 19 | 228 | 146
percent impairment
  End of treatment: number analyzed (Participants) | 19 | 226 | 140
  End of treatment | 0.0 [-10.0 to 10.0] | 0.0 [-20.0 to 0.0] | 0.0 [-10.0 to 10.0]
  12 weeks post treatment: number analyzed (Participants) | 18 | 226 | 138
  12 weeks post treatment | 0.0 [-20.0 to 0.0] | 0.0 [-20.0 to 0.0] | 0.0 [-20.0 to 0.0]
  24 weeks post treatment: number analyzed (Participants) | 18 | 223 | 135
  24 weeks post treatment | -5.0 [-30.0 to 0.0] | -10.0 [-30.0 to 0.0] | 0.0 [-30.0 to 0.0]

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after last dose. The median duration of treatment was 84 days.
Arm/Group | 2 DAA + RBV | 3 DAA Without RBV | 3 DAA + RBV
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/229 | 2/146
Serious Adverse Events (participants affected / at risk) | 3/19 | 3/229 | 8/146
Other Adverse Events (participants affected / at risk) | 8/19 | 2/229 | 26/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA + RBV (N=19) | 3 DAA Without RBV (N=229) | 3 DAA + RBV (N=146)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellullar Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA + RBV (N=19) | 3 DAA Without RBV (N=229) | 3 DAA + RBV (N=146)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 17 (17)
Asthenia (General disorders) | 1 (1) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 (4) | 1 (1) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT02640547/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT02640547/SAP_001.pdf